CLINICAL TRIAL: NCT05954325
Title: Extracorporal Apheresis Hannover Medical School Study in Post COVID-19 Patients
Brief Title: Immunoadsorption vs. Sham Treatment in Post COVID-19 Patients With Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXTINCT post COVID
Record Dates: First submitted 2023-07-19; First posted 2023-07-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Post-Acute COVID-19 Syndrome
Keywords: Post COVID syndrome; Fatigue; Immunoadsorption
MeSH Terms: conditions — Fatigue; Post-Acute COVID-19 Syndrome | interventions — Blood Component Removal

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, sham-controlled trial
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunoadsorption (Experimental): 5 immunoadsorption treatments
  Interventions: Procedure: Immunoadsorption vs. sham immunoadsorption
- Sham immunoadsorption (Sham Comparator): 5 sham immunoadsorption treatments
  Interventions: Procedure: Immunoadsorption vs. sham immunoadsorption

INTERVENTIONS:
Procedure: Immunoadsorption vs. sham immunoadsorption — 5 treatments within 14 days
  Other Names: Apheresis

SUMMARY:
The complex clinical symptoms of post COVID syndrome, especially chronic fatigue, pose a major challenge to patients and to the health care system and are frequently refractory to therapeutic intervention. There is increasing evidence that a dysregulated post-viral immune response may be involved in the pathogenesis of post COVID syndrome. In uncontrolled case studies, an improvement of fatigue symptoms after removing autoantibodies has been reported in post COVID patients. However, there is a lack of prospective, sham controlled studies. We initiate an interventional, randomised, sham treatment-controlled prospective study, the EXTINCT post COVID study, which aims to scientifically test the therapeutic efficacy of an extracorporeal apheresis procedure (immunoadsorption) for the treatment of a well characterized cohort of patients with post COVID syndrome, while at the same time providing basic research evidence for an understanding of the pathogenesis of post COVID syndrome. Thereby, we expect to obtain important insights into the diagnosis, treatment and pathophysiology of post-COVID syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Chronic Fatigue Syndrome (CFS) according to Canadian Consensus Criteria (at two time points > 4 weeks apart) with a duration of > 6 months with new onset < 12 weeks after PCR test confirmed SARS-CoV2-infection
3. Chalder Fatigue Scale >/= 4 binary scale (at two time points > 4 weeks apart)
4. Post exertional malaise >/= 14 h (at two time points > 4 weeks apart)
5. Bell Scale 20-50 (at two time points > 4 weeks apart)
6. Willing to comply with all aspects of the protocol, including blood draws, magnetic resonance imaging and ophthalmological evaluation
7. Patient is able to understand and fully participate in the activities of the study and consent in accordance with guidelines
8. Female patients of childbearing potential who are sexually active must be willing to use an acceptable form of contraception. Female patients must not be pregnant, planning to become pregnant, or be actively breastfeeding through the entire period.

Exclusion citeria:

1. Chronic fatigue due to other medical or psychological condition
2. Preexisting chronic fatigue prior to COVID infection
3. Oxygen requirement or ventilation during acute phase of COVID
4. Positive SARS-CoV-2-PCR test at the beginning of the study
5. Comorbidity bearing risk that patient might not tolerate treatment as judged by investigator including among others: malignant disease within the last 5 years, moderate to severe renal impairment (eGFR <60 ml/min), cardiac insufficiency (LVEF <40%), severe coronary heart disease, severe hypercoagulability
6. Acute or severe psychiatric disease
7. Active/acute infectious diseases like CMV, EBV, HBV, HCV, HIV, TBC
8. Patients who in the investigator's opinion might not be suitable for study (difficult peripheral venous access, not able to complete questionnaires e.g. due to language problems)
9. Taking immunosuppressive medication >3 weeks within 12 months before study inclusion
10. Any apheresis therapy before study inclusion
11. Contraindications for magnetic resonance imaging
12. Patients revealing abnormal brain structures visible in MR images
13. Patients with pre-existing ophthalmological condition or diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Chalder Fatigue Scale | 12 weeks
  Time course of fatigue symptoms as determined based on Chalder Fatigue Scale (ranging from 0 to 33), higher values indicating a higher burden of fatigue symptoms

SECONDARY OUTCOMES:
Cognitive Function | 12 weeks
  Assessment of cognitive function measured by Montreal Cognitive Assessment (Scale 0-30), lower values indicating cognitive impairment
Post exertional malaise symptoms | 12 weeks
  Assessment of frequency and severity of post exertional malaise symptoms (frequency: 0-20, severity: 0-20, duration), higher values indicating a higher burden of post exertional malaise symptoms
Measure of health status | 12 weeks
  Evaluation of health status by Short Form Health Survey (SF-36)
Depression and Anxiety | 12 weeks
  Symptoms of depression and anxiety measured by Hospital Anxiety and Depression Scale (HADS)
Autonomic dysfunction | 12 weeks
  Symptoms of autonomic dysfunction assessed by Composite Autonomic Symptom Score (COMPASS 31), generating a weighted score from 0 to 100, with higher scores representing higher symptom burden
6-min. walk test | 12 weeks
  Walking distance, oxygen saturation, heart rate and dyspnea assessed during 6-min. walk test
Hand grip strength | 12 weeks
  Hand grip strength measured via digital hand dynamometer
Optical coherence tomography angiography | 12 weeks
  Assessment of retinal microcirculation
Cranial magnetic resonance imaging and spectroscopy | 12 weeks
  Cranial magnetic resonance imaging and assessment of region-dependent metabolic distributions
Symptoms related to chronic fatigue before and after immunoadsorption | 12 weeks
  Change of symptoms as measured by Fluge score, using a scale ranging from 1 to 10 (higher values representing higher symptom load) assessing 32 fatigue related symptoms and their intra-patient change from baseline to follow-up
Neurocognitive function | 12 weeks
  Attentional deficits as assessed by Test of Attentional Performance

OTHER OUTCOMES:
Safety and tolerability of immunoadsorption treatment | 12 weeks
  Number of treatment emergent adverse events, serious adverse events and discontinuation due to treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Goedecke, MD, Principal Investigator — Hannover Medical School, Department of Nephrology and Hypertension
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No